CLINICAL TRIAL: NCT00510107
Title: A Randomized Phase II Trial of Weekly Docetaxel/Cisplatin Versus Weekly Docetaxel/Oxaliplatin in Previously Untreated Patients With Advanced Gastric Cancer
Brief Title: Weekly Docetaxel Plus Cisplatin or Oxaliplatin for AGC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gachon University Gil Medical Center (Other)
Collaborators: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMO-GI-72
Record Dates: First submitted 2007-07-31; First posted 2007-08-01 (Estimated); Last update posted 2007-08-01 (Estimated); Status verified 2007-07

CONDITIONS: Stomach Neoplasm; Stage IV; Recurrent
MeSH Terms: conditions — Stomach Neoplasms; Recurrence | interventions — Oxaliplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Docetaxel 35 mg/m2 will be administered on days 1 and 8. Cisplatin 60 mg/m2 will be administered on day 1 every 3 weeks.
  Interventions: Drug: Cisplatin
- 2 (Experimental): Docetaxel 35 mg/m2 will be administered on days 1 and 8. Oxaliplatin 120 mg/m2 will be administered on day 1 every 3 weeks.
  Interventions: Drug: oxaliplatin

INTERVENTIONS:
Drug: oxaliplatin — oxaliplatin 120 mg/m2 will be given on day 1.
  Other Names: Eloxatin
  Arms: 2
Drug: Cisplatin — Cisplatin 60 mg/m2 will be given on day 1.
  Arms: 1

SUMMARY:
To evaluate the efficacy and safety of weekly administered combination of docetaxel/cisplatin and docetaxel/oxaliplatin in chemotherapy-naïve patients with advanced gastric cancer. The primary endpoint will be the response rate.

DETAILED DESCRIPTION:
Gastric cancer is the most frequently occurring malignancy in Korea, and is one of the main causes of cancer death. While treatment options for AGC have expanded in recent years to include newer agents such as taxanes, irinotecan and oxaliplatin, myelosuppression remains a problem. Recently, weekly schedule of docetaxel is appealing due to limited incidence of severe myelosuppression compared with standard 3-weekly regimen. This altered toxicity profile suggests a potential for better tolerance and increased dose intensity.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven gastric cancer
* aged 75 years or less
* performance status 0 to 2
* no prior chemotherapy
* inoperable, recurrent, or metastatic
* normal marrow, hepatic and renal functions

Exclusion Criteria:

* active infections
* severe co-morbidities
* pregnant or lactating women
* active brain metastasis
* neuropathy of grade 2 or higher

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2007-07; Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
response rate

SECONDARY OUTCOMES:
safety

CONTACTS AND LOCATIONS:
Overall Officials: Se Hoon Park, MD, Principal Investigator — Gachon University Gil Medical Center, Incheon, Korea
Locations (1):
- Gachon University Gil Medical Center, Incheon, Incheon, South Korea